CLINICAL TRIAL: NCT06233019
Title: Efficacy of Glycolic Acid 15%Plus Salicylic Acid 2% Gel in Treatment of Plane Wart
Brief Title: Glycolic Acid Plus Salicylic Acid in Treatment of Plane Wart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Abo Elmagd Abd El Razak, Resident of Dermatology, Andrology and Venereology in Nag Hammadi General Hospirtal (Qena), Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: glycolicandsalicylicacidinwart
Record Dates: First submitted 2023-11-21; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-11

CONDITIONS: Plane Wart
Keywords: glycolic acid-Salicylic Acid-Treatment of Plane Wart
MeSH Terms: interventions — glycolic acid; Salicylic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- efficacy of glycolic acid 15%plus salicylic acid 2% gel in treatment of Plane wart . (Other)
  Interventions: Other: Glycolic Acid Plus Salicylic Acid in Treatment of Plane Wart

INTERVENTIONS:
Other: Glycolic Acid Plus Salicylic Acid in Treatment of Plane Wart — Prior to the procedure, patients will be instructed to avoid sun exposure during the treatment and to use broad spectrum sunscreen The treatment was started once daily over the entire face and maintained for two months. A fine layer of Glycolic Acid Plus Salicylic Acid face gel was applied on the whole surface where the warts were present, avoiding the eyelids and lips. In children 7 to 10 years of age, face gel was applied by their parents. Clinical controls were performed at Weeks 2, 4, 6, and 8.

SUMMARY:
To determine clinical efficacy of glycolic acid 15%plus salicylic acid 2% gel in treatment of Plane wart .

DETAILED DESCRIPTION:
Warts are typically small, rough, hard growths that are similar in color to the rest of the skin. They typically asymptomatic , except when on the bottom of the feet, where they may be painful While they usually occur on the hands and feet, they can also affect other locations One or many warts may appear They are not cancerous .

Warts are caused by infection with human papillomavirus(HPV). Factors that increase the risk include use of public showers, working with meat, eczema and a weak immune system. The virus is believed to enter the body through skin that has been damaged slightly.

Warts are classified to common wart, plane wart, plantar wart, genital wart. Plane warts are circumscribed papules with hyperkeratotic surfaces that can occur singly or in groups. In these types of warts, the human papilloma virus (HPV) has been shown to infect the keratinocyte. Although no viral subtype is absolute, typically the infection is with HPV types 3, 10, 28, and 41 These warts are small in size (1-5mm), flat, or slightly elevated lesions. Plane viral warts typically present as skin-colored or light brownish,papules on the face, beard area, or on the back of the hands, and primarily affect children.

Plane warts can greatly affect a patient's quality of life, and their persistence or recurrence cause frustration.

Their evolution is variable, and although two thirds of cases regress spontaneously in the course of two years due to immunological mechanism

The following therapies have been used in the treatment of Plane wart with varying success: salicylic acid, cryotherapy, retinoic acid, photodynamic therapy (topical 5-aminolevulinic acid photodynamic therapy), pulsed dye laser (PDL), and Candida antigen.

New medication is a combination of glycolic acid 15% plus salicylic acid 2% gel.

Glycolic acid has been used in the treatment of Plane wart . It has been suggested that alpha-hydroxy acids can produce an authentic exfoliation and dehiscence of the coenocytes from recently formed layers of the stratum corneum. Alpha-hydroxy acids also reduce the number of desmosomes and tonofilaments.in this study all patients will be instructed to avoid sun exposure during the treatment and to use broad spectrum sunscreen The treatment was started once daily over the entire face and maintained for two months. A fine layer of face gel was applied on the whole surface where the warts were present, avoiding the eyelids and lips. In children 7 to 10 years of age, face gel was applied by their parents. Clinical controls were performed at Weeks 2, 4, 6, and 8.

ELIGIBILITY:
Inclusion criteria Site: face

Exclusion criteria :

1. Photosensitivity
2. Scaring keloid
3. Herpes simplex
4. Pregnancy & Lactation

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
treatment of plane wart | 8weeks
  Evaluation of the efficacy of topical glycolic acid plus salicylic acid in treatment of plane wart.
  Response to treatment will be evaluated by the decrease in number or size of plane wart.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Result] Rodriguez-Cerdeira C, Sanchez-Blanco E. Glycolic acid 15% plus salicylic acid 2%: a new therapeutic pearl for facial flat warts. J Clin Aesthet Dermatol. 2011 Sep;4(9):62-4. PMID 21938272